CLINICAL TRIAL: NCT01744769
Title: Effects of Thyroid Hormone Withdrawal on Metabolic and Cardiovascular Parameters During Radioactive Iodine Therapy in Differentiated Thyroid Cancer
Brief Title: Effects of Thyroid Hormone Withdrawal on Metabolic Parameters During Radioactive Iodine Therapy in Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Suk Kyeong Kim, Associate professor, Konkuk University Medical Center
Other Study IDs: KUH1010379
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Hypothyroidism
Keywords: thyroid cancer; hypothyroidism; metabolic parameters; Hypothyroidism after levothyroxine withdrawal
MeSH Terms: conditions — Hypothyroidism; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypothyroidism for RAI: The group of patients who experience hypothyroidism after thyroid hormone withdrawal for radioactive iodine(RAI) therapy

SUMMARY:
1. The incidence of differentiated thyroid cancer is increasing in Korea. A significant number of them experience severe hypothyroidism in preparation for radioactive iodine (RAI) therapy after total thyroidectomy.
2. Because the function of thyroid hormone is closely linked with lipid and glucose metabolism, overt hypothyroidism after thyroid hormone withdrawal during RAI therapy may induce the changes of metabolic parameters.
3. We investigate the effects of thyroid hormone withdrawal on metabolic and cardiovascular parameters during radioactive iodine therapy in differentiated thyroid cancer.

DETAILED DESCRIPTION:
1. Study design measurement of various parameters during hypothyroid state (before 1 month, the day and after 1 month of RAI therapy)
2. Measurements

   1. Measurement of metabolic and cardiovascular parameters

      * glucose profiles : HbA1c, fasting glucose level
      * lipid profiles : free fatty acid, total, LDL-, HDL-, cholesterol, triglyceride
      * adipocytokines : retinol binding protein(RBP)
      * 4, leptin, resistin, adiponectin
      * markers of endothelial and cardiac function : high-sensitivity C-reactive protein(hsCRP), homocystein, B-type natriuretic peptide(BNP)
      * bone turnover markers : CTX, bone ALP
   2. Scoring of symptoms and signs of hypothyroidism (Zulewski score)

      * symptoms
      * physical signs

ELIGIBILITY:
Inclusion Criteria:

* radioiodine therapy after total thyroidectomy in differentiated thyroid cancer
* age over 18

Exclusion Criteria:

* kidney failure, liver failure, heart failure
* infection
* inflammation
* autoimmune disease
* other chronic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who experience severe hypothyroidism after thyroid hormone withdrawal for radioiodine therapy in differentiated thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Changes of metabolic parameters | Before 1month of radioiodine therapy, Day of radioiodine therapy, After 1 month of radioiodine therapy
  * glucose profiles : HbA1c, fasting glucose level
  * lipid profiles : free fatty acid, total, LDL-, HDL-, cholesterol, triglyceride
  * adipocytokines : retinol binding protein(RBP)4, leptin, resistin, adiponectin
  * markers of endothelial and cardiac function : high-sensitivity C-reactive - protein(hsCRP), homocystein, B-type natriuretic peptide(BNP)

SECONDARY OUTCOMES:
Changes of bone turnover markers | Before 1month of radioiodine therapy, Day of radioiodine therapy, After 1 month of radioiodine terapy
  * bone formation marker: bone ALP
  * bone resorption marker: CTX

CONTACTS AND LOCATIONS:
Overall Officials: Suk Kyeong Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea